CLINICAL TRIAL: NCT04540887
Title: Investigation of Potential Therapeutic Effects of Pulsed Electromagnetic Field for the Treatment of Symptoms Associated With Interstitial Cystitis/Bladder Pain Syndrome
Brief Title: PEMF Therapy to Treat Interstitial Cystitis/Bladder Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00068066
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Results first posted 2022-07-20 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2021-07

CONDITIONS: Interstitial Cystitis; Chronic Interstitial Cystitis; Bladder Pain Syndrome
Keywords: Interstitial Cystitis; Bladder Pain Syndrome; Painful Bladder Syndrome; IC; BPS; Painful Bladder; Urinary urgency; Urinary frequency; Nocturia; Urinary incontinence
MeSH Terms: conditions — Cystitis, Interstitial; Nocturia; Urinary Incontinence | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a single center clinical series evaluating symptom relief following a 4-week trial of PEMF therapy. From our registry of IC/BPS patients at Wake Forest Baptist Health Urology we will recruit women, ages 18-80, who have met all inclusion and exclusion criteria. Upon enrollment, each participant will be taught how to administer home treatment with the Bio Electro Magnetic Energy Regulation (BEMER) PEMF devices which consist of a total body mat (B.Body) plus a targeted pelvic mat (B.Pad) and control unit. Following the brief in-clinic training, participants will be sent home with the PEMF devices (preset to deliver the same level of energy every time) and self-administer therapy sessions, twice daily (once in the morning, once in the evening) for 8 minutes at a time. Participants will complete questionnaires as well as keep a 3-day voiding diary to record any changes in IC/BPS symptoms/pain at enrollment, 4 weeks after using PEMF therapy, and 12 weeks post-enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): Treatment will be provided via self-administration of pulsed electromagnetic field (PEMF) therapy using the B. Body (whole body mat), B. Pad (targeted pelvic mat), and Control Unit. The participant will lay the B. Body mat on any flat surface (i.e. floor, bed, reclining chair, etc.) and lie down on the mat with the smaller B. Pad placed directly over their pelvic area. Then, the participant will turn the PEMF device on using the attached control unit, which has been pre-programmed to deliver the same level of energy every time. Participants will be instructed to administer this home treatment twice a day (morning and evening) for 8-minute sessions over a four-week period. As this is a single-group assignment, all participants will be given the PEMF device.
  Interventions: Device: Pulsed Electromagnetic Field (PEMF) Therapy

INTERVENTIONS:
Device: Pulsed Electromagnetic Field (PEMF) Therapy — PEMF therapy will be self-administered by all trial participants using the B. Body, B. Pad, and Control Unit. Participants will administer this therapy twice a day (morning and evening) for 8-minute sessions over a four week period.
  Other Names: BEMER B. Body; BEMER B. Pad; BEMER Control Unit

SUMMARY:
The purpose of this study is to gather information from the investigation of a non-pharmacological (non-drug) treatment known as low frequency pulsed electromagnetic field (PEMF). The study team will be distributing the PEMF therapy to female subjects with Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS) to measure its ability to decrease pelvic pain. The results, from multiple questionnaires and voiding diaries, will be compared when participants are enrolled for treatment, at 4 weeks after using PEMF therapy, and 12 weeks post-enrollment.

DETAILED DESCRIPTION:
Interstitial cystitis/bladder pain syndrome (IC/BPS) is a clinical diagnosis based primarily on chronic symptoms of pain perceived by the patient to emanate from the bladder and/or pelvis associated with urinary urgency or frequency in the absence of another identified cause for the symptoms. Although it is not a life-threatening disease, the chronicity and severity of pain, along with urinary symptoms, causes great impairment in a patient's quality of life. IC/BPS poses as a significant clinical challenge for many reasons. For one, the pathophysiology described in the literature is incompletely determined and likely multi-factorial, including factors such as inflammation, neurovascular dysfunction, ion imbalance, and impaired urothelial cell integrity. Consequently, there are many options for IC/BPS therapy, many of which are driven primarily by patient-reported symptoms. In this regard, IC/BPS patients with moderate to severe pain typically require multi-modal therapy, often resulting in incomplete or no resolution of symptoms. Another clinical challenge is the heterogeneity of the symptoms. While pelvic pain is the distinguishing characteristic, patients with IC/BPS also routinely present with additional urological and non-urological medical symptoms and syndromes. This has led to the description of two specific sub-phenotypes in IC/BPS based on anesthetized bladder capacity (BC), in which patients with BC < 400 cc are more likely to experience severe pain, urgency and frequency (bladder centric sub-phenotype), and patients with BC > 400 cc (non-bladder centric sub-phenotype) have a higher prevalence of non-urological associated syndromes (NUAS) such as fibromyalgia, chronic fatigue symptoms, irritable bowel syndrome, endometriosis and sicca syndrome.

Pulsed Electromagnetic Field (PEMF) therapy may present a promising alternative therapy for IC/BPS. PEMF is a safe, non-invasive, and effective therapy currently used for wound healing, bone-related diseases (osteoarthritis, RA), and chronic pain states (chronic lower back pain, fibromyalgia), the latter of which is frequently associated with IC/BPS as NUAS. Based on Faraday's law, electromagnetic interactions (e.g. PEMF) with biological processes and conditions (e.g. IC/BPS) will theoretically address many of the proposed pathophysiological causes of the condition. While the mechanism(s) of action are not fully understood, PEMF therapy has been shown in several studies (randomized, double-blinded, placebo-controlled trials) to decrease the output of pro-inflammatory proteins, improve oxygenation of blood and tissue, stabilize transmembrane action potential and ion channels, and stimulate tissue regeneration. Thus, PEMF may provide a safe, non-invasive therapeutic option that would be complementary to, or serve as an alternative for, the treatments that are currently being administered in IC/BPS for pain reduction. Of note, PEMF has demonstrated an excellent safety profile with no associated systemic risks reported to date. Additionally, the application of exogenous PEMF to stimulate the pelvic floor muscle has recently been introduced for treating urge and/or stress urinary incontinence and overactive bladder. Furthermore, if patient safety and efficacy for pain reduction are demonstrated, these feasibility studies will provide the foundation for larger multi-site trials to determine additional parameters regarding the appropriate number of treatments as well as the duration of benefit (pain relief) following treatments.The purpose of this study will be to determine if PEMF therapy in patients with IC/BPS is an effective treatment in reducing pelvic pain.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between 18 and 80 years old
* Participants must have already been diagnosed with interstitial cystitis/bladder pain syndrome
* Subjects must have a bladder capacity greater than 400 cc
* Participants must have scored at least a 6 or higher on Numeric Rating Scale questionnaire
* Participants must not have any cognitive disabilities
* Participants must not have taken any narcotic medication for at least three months before being enrolled in this clinical trial

Exclusion Criteria:

* Participants must not have any history of bladder, uterine, ovarian, or vaginal cancer, urethral diverticulum, spinal cord injury, stroke, Parkinson's disease, multiple sclerosis, spina bifida, radiation cystitis, cyclophosphamide treatment, or genital herpes
* Patients cannot have an implanted pace-maker or metal prosthesis
* Participants cannot have a urinary tract infection at the time of enrollment or be currently pregnant
* Patients must not have a body mass index greater than 40

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Walker, PhD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van de Merwe JP, Nordling J, Bouchelouche P, Bouchelouche K, Cervigni M, Daha LK, Elneil S, Fall M, Hohlbrugger G, Irwin P, Mortensen S, van Ophoven A, Osborne JL, Peeker R, Richter B, Riedl C, Sairanen J, Tinzl M, Wyndaele JJ. Diagnostic criteria, classification, and nomenclature for painful bladder syndrome/interstitial cystitis: an ESSIC proposal. Eur Urol. 2008 Jan;53(1):60-7. doi: 10.1016/j.eururo.2007.09.019. Epub 2007 Sep 20. PMID 17900797
- [Background] Vasudevan V, Moldwin R. Addressing quality of life in the patient with interstitial cystitis/bladder pain syndrome. Asian J Urol. 2017 Jan;4(1):50-54. doi: 10.1016/j.ajur.2016.08.014. Epub 2016 Dec 2. PMID 29264207
- [Background] Keay SK, Birder LA, Chai TC. Evidence for bladder urothelial pathophysiology in functional bladder disorders. Biomed Res Int. 2014;2014:865463. doi: 10.1155/2014/865463. Epub 2014 May 8. PMID 24900993
- [Background] Parsons CL. The role of a leaky epithelium and potassium in the generation of bladder symptoms in interstitial cystitis/overactive bladder, urethral syndrome, prostatitis and gynaecological chronic pelvic pain. BJU Int. 2011 Feb;107(3):370-5. doi: 10.1111/j.1464-410X.2010.09843.x. Epub 2010 Dec 22. PMID 21176078
- [Background] Christmas TJ, Rode J, Chapple CR, Milroy EJ, Turner-Warwick RT. Nerve fibre proliferation in interstitial cystitis. Virchows Arch A Pathol Anat Histopathol. 1990;416(5):447-51. doi: 10.1007/BF01605152. PMID 2107633

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral from the existing database of patients with interstitial cystitis seen at Wake Forest Baptist Health Urology between February 2021 and November 2021. One participant was identified and enrolled via direct communication with investigators based on information found on clinicaltrials.gov.
Pre-assignment Details: Of 10 enrolled participants, 10 were successfully screened and met all inclusion criteria. However, 2 of the 10 participants experienced exigent personal circumstances and voluntarily withdrew from the study before their 4-week follow-up visit. These participants were subsequently excluded from data analysis.
Groups:
- Pulsed Electromagnetic Field Therapy (PEMF): Treatment will be provided via self-administration of pulsed electromagnetic field (PEMF) therapy using the B. Body (whole body mat), B. Pad (targeted pelvic mat), and Control Unit. The participant will lay the B. Body mat on any flat surface (i.e. floor, bed, fully reclined chair, etc.) and lie down on the mat with their spine straight and the smaller B. Pad straddled between their legs with the coils placed directly over the pelvic area. The participant will then turn the PEMF device on using the attached control unit, which has been pre-programmed to deliver the same amount and intensity of energy every time. Participants will be instructed to administer this home treatment twice a day (morning and evening) for 8-minute sessions over a four-week period. As this is a single-group assignment, all participants will be given the PEMF device.
Period: Overall Study
Arm/Group | Pulsed Electromagnetic Field Therapy (PEMF)
Started | 10
Completed | 8
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pulsed Electromagnetic Field Therapy (PEMF)
Number analyzed (Participants) | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [47.75 to 60.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Numeric Rating Scale (NRS) Score [Mean (Standard Deviation); unit: units on a scale] | 6.875 (0.641)
Length of IC/BPS Diagnosis [Mean (Standard Deviation); unit: years] | 10.7 (5.335)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.34 (6.507)

OUTCOME MEASURES:

1. Primary Outcome: Pelvic Pain, as Measured by the Numeric Rating Scale (NRS)
Description: The NRS evaluates average pain intensity. It appears as a horizontal line with an eleven-point range. The NRS is labeled from 0 to 10, with 0 indicating no pain and 10 indicating severe pain ("worst pain imaginable").
Time Frame: Baseline before beginning treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pulsed Electromagnetic Field Therapy (PEMF)
Number analyzed (Participants) | 10
score on a scale | 6.70 (0.675)

2. Primary Outcome: Change From Baseline Pelvic Pain, as Measured by the Numeric Rating Scale (NRS)
Description: as for outcome 1
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pulsed Electromagnetic Field Therapy (PEMF)
Number analyzed (Participants) | 8
score on a scale | 4.18 (1.462)

3. Primary Outcome: Change From Baseline Pelvic Pain, as Measured by the Numeric Rating Scale (NRS)
Description: as for outcome 1
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pulsed Electromagnetic Field Therapy (PEMF)
Number analyzed (Participants) | 8
score on a scale | 5.34 (1.845)

4. Secondary Outcome: Change in IC/BPS Symptoms, as Measured by O'Leary-Sant Interstitial Cystitis Problem Index (ICPI)
Description: The ICPI (score range: 0-16 points) contain four questions related to urinary and pain symptoms. For the problem index, all four questions utilize a range of 0-4 with 0 indicating it is no problem and 4 indicating it is a big problem. Higher scores indicate more severe symptoms and greater disease progression, while lower scores indicate less severe symptoms and less disease progression.
Time Frame: Baseline before beginning treatment, Week 4, and Week 12
Population: Of 10 participants initially enrolled, 2 experienced exigent personal circumstances and voluntarily withdrew from the study. These participants were included in the baseline data analysis but were excluded from the 4- and 8-week post-enrollment data analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pulsed Electromagnetic Field Therapy (PEMF)
Number analyzed (Participants) | 10
scores on a scale
  Baseline | 13 (1.927)
  Week 4: number analyzed (Participants) | 8
  Week 4 | 9.125 (4.581)
  Week 12: number analyzed (Participants) | 8
  Week 12 | 10.75 (3.742)

5. Secondary Outcome: Change in IC/BPS Symptoms, as Measured by Wake Forest Baptist Health IC/BPS Global Response Assessment (GRA)
Description: The GRA asks participants to list any in-office treatments, home treatments, medications, or procedures they have had in the past year for IC/BPS. Then, they are asked to score those treatments based on a seven point scale (-3 to +3) with -3 indicating their symptoms became markedly worse and +3 indicating their symptoms were markedly improved after treatment.
Time Frame: Baseline, 4-weeks post-treatment, and 8-weeks post-treatment
Population: Of 10 participants initially enrolled, 2 experienced exigent personal circumstances and voluntarily withdrew from the study. These participants were included in the baseline data analysis but were excluded from the 4- and 8-week post-enrollment data analysis. Additionally, 1 patient at the 4-week post-treatment evaluation and 3 patients in the 8-week post-treatment evaluation did not specifically list PEMF therapy in the GRA, and therefore their data were excluded from analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 10
score on a scale
  Baseline | 0 [0 to 0]
  4-weeks post-treatment: number analyzed (Participants) | 7
  4-weeks post-treatment | 2 [1 to 2]
  8-weeks post-treatment: number analyzed (Participants) | 5
  8-weeks post-treatment | 2 [1 to 3]

6. Secondary Outcome: Change in IC/BPS Symptoms, as Measured by O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI)
Description: The ICSI (score range: 0-19 points) contains four questions related to urinary and pain symptoms. For the symptoms index, 3 of the 4 questions utilize a range of 0-5 with 0 indicated the symptom is never experienced and 5 indicating the symptom is almost always experienced. The fourth question utilizes a range of 0-4 with 0 indicating the symptom is never experienced and 4 indicating the symptom is almost always experienced. Higher scores indicate more severe symptoms and greater acuity of disease progression, while lower scores indicate less severe symptoms and lower acuity of disease progression.
Time Frame: Baseline before beginning treatment, Week 4, and Week 12
Population: Of 10 participants initially enrolled, 2 experienced exigent personal circumstances and voluntarily withdrew from the study. These participants were included in the baseline data analysis but were excluded from Week 4 and Week 12 data analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 10
scores on a scale
  Baseline before beginning treatment | 13.875 (2.949)
  Week 4: number analyzed (Participants) | 8
  Week 4 | 9 (4.781)
  Week 12: number analyzed (Participants) | 8
  Week 12 | 10 (3.741)

7. Secondary Outcome: Change in IC/BPS Symptoms, as Recorded in Patient Voiding Diary - Void and Intake Measurements
Description: Participants will be instructed on how to complete 3-day voiding diary prior to initial office visit and following assessments. The participant will use a new diary sheet for every 24-hour period. Data analysis will be measured based on urgency score, total urine volume (TUV) (mL), maximum voided volume (MVV) (mL), mean voided volume (mL), and fluid intake (mL).
  For TUV, MVV, and mean voided volume, higher voided volume (in mL) indicates more efficient bladder-emptying and less severe symptoms, while a lower voided volume (in mL) indicates less efficient bladder-emptying and more severe symptoms.
Time Frame: Baseline before beginning treatment and Week 4
Population: Of 10 participants enrolled, 2 experienced exigent personal circumstances and voluntarily withdrew from the study. Their data was excluded from data analysis. Additionally, of the remaining 8 participants, 2 failed to complete their voiding diaries in its entirety and one additional participant did not complete her fluid intake. Thus, 6 women had evaluable voiding information and 5 had data for fluid intake to evaluate.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Treatment
Number analyzed (Participants) | 10
mL
  Total Urine Volume (TUV in mL) (Baseline): number analyzed (Participants) | 6
  Total Urine Volume (TUV in mL) (Baseline) | 2808.68 (1498.93)
  Total Urine Volume (TUV in mL) (Week 4): number analyzed (Participants) | 6
  Total Urine Volume (TUV in mL) (Week 4) | 2511.67 (1514.67)
  Maximum Voided Volume (MVV in mL) (Baseline): number analyzed (Participants) | 6
  Maximum Voided Volume (MVV in mL) (Baseline) | 406.71 (234.13)
  Maximum Voided Volume (MVV in mL) (Week 4): number analyzed (Participants) | 6
  Maximum Voided Volume (MVV in mL) (Week 4) | 454.29 (307.60)
  Mean Voided Volume (mL) (Baseline): number analyzed (Participants) | 6
  Mean Voided Volume (mL) (Baseline) | 215.45 (116.38)
  Mean Voided Volume (mL) (Week 4): number analyzed (Participants) | 6
  Mean Voided Volume (mL) (Week 4) | 229.67 (140.63)
  Fluid Intake (Baseline): number analyzed (Participants) | 5
  Fluid Intake (Baseline) | 1701.52 (600.00)
  Fluid Intake (Week 4) | 1594.69 (668.17)

8. Secondary Outcome: Change in IC/BPS Symptoms, as Recorded in Patient Voiding Diary - Number of Voids
Description: Participants will be instructed on how to complete 3-day voiding diary prior to initial office visit and following assessments. The participant will use a new diary sheet for every 24-hour period with sections identifying time of day (with wake time and bed time indicated by participant), fluid intake (type of fluid ingested and amount in oz), urination (amount in oz voided into urinary hat or urinal), amount of urine drained via catheter if applicable, leaks (any time participant experienced involuntary urine loss indicated by a check mark in the corresponding time column) if applicable, and pad changes if applicable. Data analysis will be measured based on daily number of voids (voids).
  For number of voids specifically, a greater number of voids in a 24-hour period indicates increased urinary frequency and more severe symptoms, while a fewer number of voids in a 24-hour period indicates decreased urinary frequency and less severe symptoms.
Time Frame: Baseline before beginning treatment and Week 4
Population: Of 10 participants enrolled, 2 experienced exigent personal circumstances and voluntarily withdrew from the study. Their data was excluded from data analysis. Additionally, of the remaining 8 participants, 2 failed to complete their voiding diaries in its entirety.
Measure: Mean (Standard Deviation); unit: voids
Arm/Group | Treatment
Number analyzed (Participants) | 10
voids
  Daily Number of Voids (Baseline): number analyzed (Participants) | 6
  Daily Number of Voids (Baseline) | 13.79 (3.33)
  Daily Number of Voids (Week 4) | 11.52 (1.79)

9. Secondary Outcome: Change in IC/BPS Symptoms, as Recorded in Patient Voiding Diary - Urgency Score
Description: Participants will be instructed on how to complete 3-day voiding diary prior to initial office visit and following assessments. The participant will use a new diary sheet for every 24-hour period with sections identifying time of day (with wake time and bed time indicated by participant), fluid intake (type of fluid ingested and amount in oz), urination (amount in oz voided into urinary hat or urinal), amount of urine drained via catheter if applicable, leaks (any time participant experienced involuntary urine loss indicated by a check mark in the corresponding time column) if applicable, and pad changes if applicable. Data analysis will be measured based on urgency score (scale: 0-3, with 0 indicating no urgency and 3 indicating maximum urgency).
  For the urgency score specifically, lower scores indicate less severe urinary symptoms/urgency while higher scores indicate more severe urinary symptoms/urgency.
Time Frame: Baseline before beginning treatment and Week 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 10
Score on a scale
  Urgency Score (range from 0-4) (Baseline): number analyzed (Participants) | 8
  Urgency Score (range from 0-4) (Baseline) | 2.12 (0.70)
  Urgency Score (range from 0-4) (Week 4): number analyzed (Participants) | 8
  Urgency Score (range from 0-4) (Week 4) | 1.91 (0.586)

ADVERSE EVENTS:
Time Frame: 36 Weeks
Arm/Group | Pulsed Electromagnetic Field Therapy (PEMF)
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
The primary limitation of this pilot clinical trial was the small sample size and absence of a control group. We recognize the potential for a significant placebo effect among this patient population. Furthermore, our results are non-generalizable as we evaluated only females, and only those that were considered to have a non-bladder centric IC/BPS phenotype. To mitigate these shortcomings, the next iteration of this trial will employ a randomized, double-blind, sham-controlled study design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT04540887/Prot_SAP_003.pdf
  • Informed Consent Form (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT04540887/ICF_004.pdf